CLINICAL TRIAL: NCT06324955
Title: A Prospective Randomized Study Comparing Positive Language vs Common Language During Inhalational Induction
Brief Title: Language During Inhalational Induction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Julia Galvez-Delgado, Anesthesiologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-P00042507
Record Dates: First submitted 2024-03-08; First posted 2024-03-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Emergence Delirium; Anesthesia; Adverse Effect
Keywords: Anesthesia induction
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common/Standard Language Group (Active Comparator)
  Interventions: Behavioral: Standard/common language during induction
- Positive Language Group (Experimental)
  Interventions: Behavioral: Positive language during induction

INTERVENTIONS:
Behavioral: Standard/common language during induction — The anesthesiologist taking care of the patient will use scripted common/standard language during the induction.
  Arms: Common/Standard Language Group
Behavioral: Positive language during induction — The anesthesiologist taking care of the patient will use scripted positive language during the induction.
  Arms: Positive Language Group

SUMMARY:
The aim of this study is to compare the impact of common (standard of care) language vs positive language used by clinicians during inhalational induction of anesthesia on anxiety and negative behaviors in children. This is a prospective randomized parallel group trial. Patients will be randomized 1:1 to the common/standard language group or the positive language group.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2 (Healthy Patients)
* Non-emergent cases
* 5-10 year olds
* Patients receiving inhalational induction

Exclusion Criteria:

* Non-English speaking
* History of prior inhalational inductions
* Hearing difficulty
* Behavioral difficulty (Autism, Oppositional Defiant Disorder)
* Patients receiving premedication other than midazolam

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Induction compliance | Through Study Completion about 1 day
  Compliance of children during mask induction as measured by the Induction Compliance Checklist (ICC) from the time patient enters the operating room until loss of lid reflex

SECONDARY OUTCOMES:
Length of induction | Through Study Completion about 1 day
  Time from start of induction to loss of lid reflex
Verbal refusal of mask | Through Study Completion about 1 day
  Patient verbal expression of refusal of the mask during start of induction until loss of lid reflex

CONTACTS AND LOCATIONS:
Overall Officials: John Fiadjoe, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States